CLINICAL TRIAL: NCT01606371
Title: Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of LY2409021 After Escalating Single Oral Dose Administration in Healthy Subjects and Patients With Type 2 Diabetes Mellitus
Brief Title: A First-in-Human Study of LY2409021 in Healthy Participants and Participants With Type 2 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 10837; I1R-FW-GLBA (Other: Eli Lilly and Company)
Record Dates: First submitted 2012-05-23; First posted 2012-05-25 (Estimated); Last update posted 2012-05-25 (Estimated); Status verified 2012-05

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — adomeglivant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (11):
- Healthy-Placebo (Placebo Comparator): Placebo (capsule) administered once, orally
  Interventions: Drug: Placebo
- Healthy-2.5 mg LY2409021 (Experimental): 2.5 mg LY2409021 administered once, orally
  Interventions: Drug: LY2409021
- Healthy-10 mg LY2409021 (Experimental): 10 mg LY2409021 administered once, orally
  Interventions: Drug: LY2409021
- Healthy-30 mg LY2409021 (Experimental): 30 mg LY2409021 administered once, orally
  Interventions: Drug: LY2409021
- Healthy-100 mg LY2409021 (Experimental): 100 mg LY2409021 administered once, orally
  Interventions: Drug: LY2409021
- Healthy-250 mg LY2409021 (Experimental): 250 mg LY2409021 administered once, orally
  Interventions: Drug: LY2409021
- Healthy-500 mg LY2409021 (Experimental): 500 mg LY2409021 administered once, orally
  Interventions: Drug: LY2409021
- Diabetic-Placebo (Placebo Comparator): Placebo (capsule) administered once, orally
  Interventions: Drug: Placebo
- Diabetic-75 mg LY2409021 (Experimental): 75 mg LY2409021 administered once, orally
  Interventions: Drug: LY2409021
- Diabetic-200 mg LY2409021 (Experimental): 200 mg LY2409021 administered once, orally
  Interventions: Drug: LY2409021
- Diabetic-500 mg LY2409021 (Experimental): 500 mg LY2409021 administered once, orally
  Interventions: Drug: LY2409021

INTERVENTIONS:
Drug: Placebo — Administered orally
  Arms: Diabetic-Placebo; Healthy-Placebo
Drug: LY2409021 — Administered orally
  Arms: Diabetic-200 mg LY2409021; Diabetic-500 mg LY2409021; Diabetic-75 mg LY2409021; Healthy-10 mg LY2409021; Healthy-100 mg LY2409021; Healthy-2.5 mg LY2409021; Healthy-250 mg LY2409021; Healthy-30 mg LY2409021; Healthy-500 mg LY2409021

SUMMARY:
The main purpose of this study is to determine the safety of LY2409021 in healthy participants and participants with diabetes. The study drug is given as single oral doses. Each participant can receive up to 3 doses, with a minimum 7 day washout between dosing periods. Side effects will be documented. This study is approximately 9 weeks long, not including screening. Screening is required within 6 weeks prior to the start of the study.

ELIGIBILITY:
Inclusion Criteria:

For all participants:

* Must be either a male, or a female who cannot become pregnant, who is either healthy or have type 2 diabetes mellitus (T2DM) but not taking medication for diabetes
* Have an hemoglobin A1c (HbA1c) value of less than or equal to 10% at screening
* Have blood and urine laboratory test results that are acceptable for the study

For healthy participants:

* Have a screening body mass index (BMI) of 18.5 to 29.9 kg/m^2 inclusive
* Have a fasting blood glucose between 3.0-5.2 millimoles/liter (mmol/L) at screening
* Have plasma glucose, two hours after ingesting an oral 75 g glucose load, less than 7.8 mmol/L

For participants with type 2 diabetes mellitus (T2DM):

* Have a screening body mass index (BMI) of 18.5 to 35 kg/m^2 inclusive
* Must weigh 45 kg or more at screening
* Have a fasting blood glucose less than 11.1 mmol/L at screening
* Have plasma glucose, two hours after ingesting an oral 75 g glucose load, greater than or equal to 11.1 mmol/L

Exclusion Criteria:

For all participants:

* Have participated in a study with a new drug in the last 30 days
* Have a history of significant heart, lung, liver, kidney, stomach or brain disease, or have any medical problems which may cause an increased risk during the study
* Have hypertension requiring more than single-agent therapy, or blood pressure greater than 140/90 millimeters of mercury (mmHg) on monotherapy
* Are allergic to LY2409021 or similar drugs
* Have a regular alcohol intake greater than 21 units/week (male), or 14 units/week (female), or are unwilling to stop alcohol as required by the study restrictions (1 unit = 360 mL of beer, or 150 mL of wine, or 45 mL of spirits)
* Intend to use other over-the-counter or prescribed medicines during 7 or 14 days respectively before the study, or during the study. Medicines for high cholesterol and high blood pressure are allowed if you have diabetes.
* Have a significant blood disorder and/or donated blood (450 ml or more) in the last 3 months

For participants with T2DM:

* Have signs of having serious problems with diabetes (For example, severe eye problems, poorly healing skin)
* Have a history of being in a coma due to low blood sugar

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2007-05; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Number of participants with one or more drug related adverse events (AEs) or any serious AEs | From first dose of study drug up to discharge (at least 14 days after last dose)

SECONDARY OUTCOMES:
Pharmacokinetics: Area under the concentration curve (AUC) of LY2409021 | From each dose of study drug up to 14 days post dose
Pharmacokinetics: Maximum concentration (Cmax) of LY2409021 | From each dose of study drug up to 14 days post dose
Change in fasting blood glucose level | From each dose of study drug up to 48 hours post dose
Change in fasting insulin level | From each dose of study drug up to 48 hours post dose
Change in fasting glucagon level | From each dose of study drug up to 48 hours post dose
Change in fasting glucagon-like peptide-1 (GLP-1) level | From each dose of study drug up to 24 hours post dose
Glucose excursion after meals | 28 hours after each dose

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-45 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Singapore, Singapore

REFERENCES:
- [Derived] Kelly RP, Garhyan P, Raddad E, Fu H, Lim CN, Prince MJ, Pinaire JA, Loh MT, Deeg MA. Short-term administration of the glucagon receptor antagonist LY2409021 lowers blood glucose in healthy people and in those with type 2 diabetes. Diabetes Obes Metab. 2015 Apr;17(4):414-22. doi: 10.1111/dom.12446. Epub 2015 Mar 2. PMID 25656305